CLINICAL TRIAL: NCT00908817
Title: Triamcinolone Paste to Reduce the Incidence of Postoperative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Park Sun-Young, Soonchunhyang University, College of medicine Bucheon Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ST
Record Dates: First submitted 2009-05-21; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Tracheal Intubation
Keywords: postoperative sore throat; tracheal intubation; lubrication; triamcinolone
MeSH Terms: interventions — Triamcinolone Acetonide; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- triamcinolone (Active Comparator)
  Interventions: Drug: triamcinolone acetonide
- chlorhexidine (Placebo Comparator)
  Interventions: Drug: chlorhexidine gluconate

INTERVENTIONS:
Drug: triamcinolone acetonide — paste applied over tracheal tube for lubrication
  Arms: triamcinolone
Drug: chlorhexidine gluconate — jelly applied over tracheal tube for lubrication
  Arms: chlorhexidine

SUMMARY:
The purpose of this study is to determine whether triamcinolone paste applied over tracheal tube is effective to reduce the incidence of postoperative sore throat after tracheal intubation.

DETAILED DESCRIPTION:
Sore throat is a common postoperative complaint after tracheal intubation. When the surgical pain is well controlled, sore throat is often the predominant complaint, therefore it is important to prevent sore throat.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II, aged between 20 and 70 years
* scheduled for elective laparoscopic cholecystectomy under general anesthesia with endotracheal intubation

Exclusion Criteria:

* recent respiratory tract infection or sore throat
* who were using analgesics or steroid preoperatively
* who have risk factors for oral cavity infection
* the surgical duration < 60 minutes or > 300 minutes

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative sore throat | postoperative day 1

SECONDARY OUTCOMES:
the severity of postoperative sore throat | postoperative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University, College of medicine Bucheon Hospital, 1174 Jung-Dong, Wonmi-Gu, Bucheon-Si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park SY, Kim SH, Lee SJ, Chae WS, Jin HC, Lee JS, Kim SI, Hwang KH. Application of triamcinolone acetonide paste to the endotracheal tube reduces postoperative sore throat: a randomized controlled trial. Can J Anaesth. 2011 May;58(5):436-42. doi: 10.1007/s12630-011-9478-6. Epub 2011 Feb 26. PMID 21359615